CLINICAL TRIAL: NCT07378722
Title: Rhythmic Auditory Stimulaton Using Personalized Music Therapy in Parkinson's Disease
Acronym: RASP-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rumesa Butt (Other)
Responsible Party: Sponsor-Investigator, Rumesa Butt, principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/15/03/34
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Parkinson s Disease
Keywords: Parkinson's disease; Rhythmic auditory stimulation; Personalized music therapy; Freezing of gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A Conventional physical therapy (Active Comparator): Participants in Group A will receive conventional physical therapy for Parkinson's disease. The intervention will be delivered three times per week for eight weeks and will include warm-up activities, stretching, balance training, gait training, and lower-limb strengthening exercises. Outcomes will be assessed at baseline and after completion of the intervention period.
  Interventions: Behavioral: conventional physical therapy
- group B Rhythmic Auditory Stimulation with Personalized Music (Experimental): Participants in Group B will receive rhythmic auditory stimulation using personalized music synchronized to individual gait cadence, in addition to conventional physical therapy. The intervention will be administered three times per week for eight weeks. Conventional therapy will include warm-up exercises, stretching, balance training, gait training, and strengthening. Outcome measures will be assessed at baseline and after completion of the intervention period.
  Interventions: Behavioral: Rhythmic Auditory Stimulation (RAS)

INTERVENTIONS:
Behavioral: conventional physical therapy — GROUP A This group will receive the conventional physical therapy protocol for 8 weeks, they will receive treatment 3 times a week and the readings will be takenat baseline and at the end of 8 weeks of treatment. Total treatment sessions will be 24
  Arms: group A Conventional physical therapy
Behavioral: Rhythmic Auditory Stimulation (RAS) — Rhythmic Auditory Stimulation (RAS) will be delivered using personalized music selected according to each participant's preferred genre and synchronized to their individual walking cadence. Auditory cues will be provided through rhythmic music or a metronome embedded within the music to facilitate temporal gait regulation and motor entrainment. During gait training, participants will be instructed to synchronize their steps with the rhythmic auditory cues while walking overground.
  The RAS intervention will be administered three sessions per week for eight weeks, with each session lasting approximately 15-20 minutes and integrated into a conventional physical therapy program. The tempo of auditory cues will be adjusted progressively based on individual performance to encourage improvements in gait initiation, stride consistency, walking velocity, and reduction in freezing episodes.
  This intervention is designed to enhance gait automaticity and balance control in individuals with Parki
  Arms: group B Rhythmic Auditory Stimulation with Personalized Music

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disorder commonly associated with gait disturbances, balance impairments, and freezing of gait, which significantly increase the risk of falls and reduce functional independence. Conventional physical therapy improves mobility in individuals with PD; however, persistent gait deficits often remain. Rhythmic Auditory Stimulation (RAS) is an emerging, evidence-based intervention that uses external auditory cues to enhance gait timing, stride length, and movement initiation.

This randomized controlled trial aims to evaluate the effectiveness of rhythmic auditory stimulation using personalized music therapy combined with conventional physical therapy compared to conventional physical therapy alone in individuals with Parkinson's disease. The primary outcomes include freezing of gait, gait velocity, and balance performance. Forty-two clinically diagnosed Parkinson's disease patients will be randomly allocated into two groups. Group A will receive conventional physical therapy, while Group B will receive rhythmic auditory stimulation using personalized music in addition to conventional therapy over an 8-week intervention period.

The findings of this study may provide clinical evidence supporting the integration of personalized rhythmic auditory stimulation into rehabilitation programs for improving gait and balance in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is characterized by progressive impairments in motor control, including bradykinesia, rigidity, postural instability, and freezing of gait. Among these, freezing of gait and balance dysfunction are particularly disabling, as they interfere with safe ambulation and daily activities. Despite pharmacological management, gait and balance impairments often persist, necessitating effective rehabilitative strategies.

Rhythmic Auditory Stimulation (RAS) is a neurologic music therapy technique that provides rhythmic external cues to facilitate movement coordination through auditory-motor entrainment. Auditory cues, particularly when synchronized with an individual's natural walking cadence, have been shown to improve gait initiation, stride length, walking speed, and movement regularity in patients with Parkinson's disease. Personalized music-based RAS may further enhance adherence, motivation, and motor performance compared to non-personalized auditory cues.

This randomized controlled trial will be conducted at University of Lahore Teaching Hospital and Shadman Medical Center, Lahore, over a duration of nine months following ethical approval. A total of 42 patients diagnosed with Parkinson's disease according to Queen Square Brain Bank criteria will be recruited using a purposive sampling technique and randomly allocated into two equal groups through computer-generated randomization.

Both groups will receive treatment three times per week for eight weeks (24 sessions). Group A will undergo a conventional physical therapy program focusing on warm-up activities, stretching, balance training, gait training, and strengthening exercises. Group B will receive rhythmic auditory stimulation using personalized music synchronized to the participant's walking cadence in addition to the same conventional physical therapy protocol.

Outcome measures will be assessed at baseline and at the end of the 8-week intervention period. The primary outcome variables include freezing of gait, gait velocity, and balance management. Data will be analyzed using SPSS version 24, with appropriate parametric or non-parametric statistical tests applied based on data distribution. A p-value of ≤ 0.05 will be considered statistically significant.

This study aims to provide high-quality clinical evidence regarding the effectiveness of rhythmic auditory stimulation using personalized music therapy as an adjunct to conventional physical therapy in improving gait and balance outcomes in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* According to the Queen Square Brain Bank standard , clinical diagnosed patients of PD Both male and females ages 45-55 The mini mental state examination scale MMSE screening without severe cognitive impairment,can cooperate with this study > 23 Mild bergs balance scale BBS score (21-40 ) score

Exclusion Criteria:

* A history of neoplasms; severe cardiovascular, respiratory, visual, auditory, andmuscular-skeletal disease; other neurological conditions; and neurologic music therapy inthelast3 months.

Other disorders that could potentially influence balance and walking.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Freezing of Gait | Baseline and after 8 weeks of intervention
  Freezing of gait will be assessed using the Freezing of Gait Questionnaire (FOGQ), a validated patient-reported outcome measure designed to quantify the frequency and severity of freezing episodes during walking, turning, and gait initiation in individuals with Parkinson's disease. Higher scores indicate greater severity of freezing of gait.

SECONDARY OUTCOMES:
Balance Performance | Baseline and after 8 weeks of intervention
  Balance performance will be evaluated using the Berg Balance Scale (BBS), a standardized clinical assessment consisting of 14 functional balance tasks. Scores range from 0 to 56, with higher scores indicating better balance and postural stability in individuals with Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rumesa Aslam, MSPTN, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- Shadman Medical Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No